CLINICAL TRIAL: NCT04534257
Title: Prospective Registry to Investigate the Safety and Efficacy of the Treatment With the Selution Sirolimus Drug Coated Balloon in TASC C and D Atheroma-occlusive Infra-Inguinal Disease in Patients With Chronic Limb Threatening Ischemia From Singapore
Acronym: PRISTINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2605
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Critical Lower Limb Ischemia; Peripheral Artery Disease
Keywords: Drug-eluting balloon; Sirolimus
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Angioplasty with SELUTION Sirolimus DCB (Experimental): Subjects with infra-inguinal occlusive lesions will be treated with SELUTION Sirolimus DCB
  Interventions: Device: SELUTION Sirolimus DCB

INTERVENTIONS:
Device: SELUTION Sirolimus DCB — Suitable lesions will be treated with SELUTION Sirolimus DCB

SUMMARY:
Extensive arterial occlusion significantly reduces arterial perfusion, and may eventually lead to Critical Limb Ischemia (CLI). The pathology gives rise to symptoms such as ischemic pain, slow healing wounds at lower extremity and gangrene. It places patients with multi-segment occlusion at high risks of amputations and mortality. The treatment methods for such long occlusive lesions are limited. Traditionally, the standard of care would be surgical revascularization. This is because lesion length have been identified in several studies as an independent risk factor for the development of restenosis after angioplasty and/or stenting. However, thanks to recent advances in endovascular techniques, such as the utilization of subintimal technique for crossing long segment occlusions, it is now possible to employ endovascular techniques for suitable patients.The re-establishment of an in-line flow, even if only temporary, can allow tissue healing, which is vital in achieving limb salvage. In addition, the use of Drug Coated Balloons (DCB) can potentially reduce restenosis rate, as Sirolimus have an anti-proliferative effect.

To date, there are few studies that have evaluated the performance of DCB in lesions that are longer than 10cm. The investigators hope to evaluate the performance of the Selution DCB when used in treatment of such lesions

ELIGIBILITY:
Inclusion Criteria

1. Age of subject is > 21 years old.
2. Patient has critical limb ischemia, presenting a score from 4 to 6 following Rutherford classification
3. Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
4. Patient is willing to comply with specified follow-up evaluations at the specified times
5. Patient has a projected life expectancy of at least 12 months and has not suffered an MI within past 30 days
6. Prior to enrolment, the guidewire has crossed the target lesion

Angiographic Inclusion Criteria

1. De novo and post-PTA re-stenotic lesions located in the SFA, popliteal and/or tibial arteries suitable for endovascular therapy
2. The target lesion is located within the SFA, popliteal and/or tibial and infra-malleolar arteries
3. The length of the target lesion is > 50mm and considered as TASC C or D lesion according to the TASC II classification.
4. The target lesion has angiographic evidence of stenosis > 50% or occlusion, which has been passed with standard guidewire manipulation and pre-dilated to <30% residual stenosis using any combination of POBA, high pressure POBA, scoring balloon, or rotablator.
5. Target vessel diameter visually estimated is >1.5mm and <7 mm below the groin to the foot
6. Lesions in the treated segment may be continuous or may have gaps present between stenoses and occlusions
7. The target lesion has both patent inflow and at least one patent outflow tract extending to below the ankle. If required, the vessels of the ankle and foot should be treated with pre-dilatation and deployment of an appropriated sized balloon (i.e. smaller sized POBA or Selution study device) to establish distal flow reconstitution and adequate foot blush prior to treatment of the target tibial lesion.
8. Inflow iliac and common femoral artery lesions can be treated during the same procedure using standard angioplasty and/or approved device. These inflow lesions must be treated first prior to consideration of treatment of the BTK lesions. The patient can be enrolled if the inflow lesions are treated with good angiographic results (must have < 30% residual stenosis and no evidence of embolization)
9. There is angiographic evidence of at least one vessel-runoff through the ankle and into the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention

Exclusion Criteria:

1. Patient refusing treatment
2. Patient is permanently wheel-chair bound or bedridden
3. Presence of a stent in the target lesion that was placed during a previous procedure
4. The intervention is being performed in preparation for a planned major amputation.
5. Untreated flow-limiting inflow lesions
6. Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
7. Previous bypass surgery in the same limb
8. Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
9. Perforation at the angioplasty site evidenced by extravasation of contrast medium
10. Untreatable lesion located at the distal outflow arteries
11. Patients with uncorrected bleeding disorder
12. Aneurysm located at the level of the SFA/popliteal artery
13. Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
14. Any condition which prevents patient from complying with the study protocol or if patient has a life expectancy of <1 year.
15. Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
16. Septicaemia or bacteraemia
17. Patient has undrained pus or spreading wet gangrene in the foot that is not controlled at the time of revascularization procedure
18. Neurotrophic ulcer or heel pressure ulcer or ulcer potentially involving calcaneus (index limb)
19. episode of acute limb ischaemia within the previous 1 month
20. Use of, atherectomy or laser devices during procedure
21. Any patient considered to be hemodynamically unstable at onset of procedure
22. Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
23. The patient is currently breast-feeding, pregnant or intends to become pregnant.
24. Subject receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.) The patient should also not receive inhibitors of CYP3A (such as Itraconazole, and Erythromycin), or inducers of CYP3A (such as Rifampycin) within 90 days following the procedure.
25. Subject has tested positive for Dengue, Covid19, Ebola, SARS, or MERS. If subject becomes infected during the course of the study, the resulting outcomes data will be recorded but will not be included the analysable results from the study.
26. Patient is participating in another research study of a device, medication, biologic or other agent within 30 days which could in the opinion of the investigator affect the results of this study
27. Any patient who has received a paclitaxel coated DCB within 30 days prior to the index procedure. If the patient receives a paclitaxel DCB in a peripheral vessel during the index procedure, that patients clinical outcomes shall not be included in calculation of the primary or secondary endpoints of the study
28. Patients with lesion to be treated with residual stenosis after POBA of >30%

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events | 30 days post-index procedure
  Composite of freedom from device- and procedure-related mortality
Freedom from clinically driven target lesion revascularization | 6 months post-index procedure
  Any re-intervention performed for more than 50% diameter stenosis at target lesion after documentation of recurrent or unresolved and continuing clinical symptoms

SECONDARY OUTCOMES:
Primary patency | 6 and 12 months post-index procedure
  Absence of hemodynamically significant stenosis on duplex ultrasound at target lesion and without target lesion revascularization between time of procedure and the given follow-up
Technical Success | Immediately post-op
  Ability to cross and dilate the lesions and achieve residual angiographic stenos no greater than 30%
Freedom from clinically-drive target lesion revascularization | 12 month post-index procedure
  Repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge at respective time points
Clinical success at follow-up | 6 and 12 months post index procedure
  Improvement of Rutherford classification at all follow-up time points of one class or more as compared to the pre-procedure Rutherford classification
Wound healing | 6 months post-index procedure
  Closure of primary wound by more than 70%
Freedom from major target limb amputation | 6 and 12 months post-index procedure
Freedom from Serious Adverse Events | 1 year post-index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital; Tze Tec Chong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No